CLINICAL TRIAL: NCT02554461
Title: Optimaliseren Van Lichaams- en Bewegingsspecifieke Kenmerken Bij Volleybalspelers Met Het Oog op Het Reduceren Van Blessures
Brief Title: Optimization of Movement Patterns in Elite Volleyball Players
Status: Completed | Type: Observational
Sponsor: Prof. Dr. F. Staes (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. F. Staes, professor, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Other Study IDs: S56955
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2016-10

CONDITIONS: Optimisation of Performance and Avoidance of Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- female players: national team players
  Interventions: Other: advise for exercices given by team staff
- male players: national team players
  Interventions: Other: advise for exercices given by team staff

INTERVENTIONS:
Other: advise for exercices given by team staff — To respond to questions asked:
  it is not the investigator who decides on the intervention, but the daily team staff (e.g. trainer, coach, PT,.....). So no predetermined intervention is provided

SUMMARY:
On the basis of clinical and movement analysis records players are informed on what parameters can be optimized in order to improve their performance and avoid injuries

ELIGIBILITY:
Inclusion Criteria:

Members of national volleyball team signing informed consent

Exclusion Criteria:

No specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female national team volleyball players
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
2D and 3D joint angles of different movements together with kinetics | 1 day
  kinematics and kinetics with regard to gait, running, jumping and arm movements. This means for example joint angles (measured by 3D motion analyses data, 2D measurement data) and kinetics (joint moments, pressure plate measurements) Time frames: these data will recorded by one measurement session. For information of clinicaltrials.gov (also other outcome measures): at this point it really is an observational study. It is a kind of "service project" for an elite athletes team. Advice is provided, but not as is meant within a real clinical trial. It might evolve to such a project, but at this state it is not the case.

SECONDARY OUTCOMES:
muscle strength | 1 day
  isokinetic measurements (expressed in Nm)
muscle strength | 1 day
  isokinetic measurements (ratio agonist/antagonist as for example ratio between knee flexors/extensors) Time frames: these data will be recorded during one measurement session. This is during same session as for primary outcome measure.
joint stability | 1 day
  nominal scale (good, poor)
joint control | 1 day
  nominal scale (good, poor)
prevalence injury past | 1 day
  interview (frequency/percentage of occurrence)
prevalence injury present | 1 day
  interview (yes/no)
(segmental) length | 1 day
  Meter
weight | 1 day
  Kg
Body mass index | 1 day
  Kg/m²

CONTACTS AND LOCATIONS:
Overall Officials: Filip f Staes, prof, Principal Investigator — UZLeuven - KU Leuven
Locations (1):
- KU Leuven/UZLeuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No